CLINICAL TRIAL: NCT02843633
Title: A Prospective Study of the BioFreedom™ Biolimus A9™ Drug Coated Stent in Patients at High Risk for Bleeding
Brief Title: LEADERS FREE II: BioFreedom™ Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16US01
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Acute Coronary Syndrome; High Bleeding Risk
Keywords: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Drug Coated Stent; Drug Eluting Stent
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Angioplasty, Balloon; Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- BioFreedom™ Drug Coated Stent (Experimental)
  Interventions: Device: BioFreedom™ Drug Coated Coronary Stent System; Drug: Antiplatelet Drug

INTERVENTIONS:
Device: BioFreedom™ Drug Coated Coronary Stent System — a non-surgical procedure that uses a catheter to place a stent to open up coronary arteries that have been narrowed by atherosclerosis
  Other Names: Coronary Angioplasty
Drug: Antiplatelet Drug — Dual antiplatelet therapy for one month followed by single antiplatelet therapy indefinitely. Aspirin and clopidogrel (or other P2Y12 inhibitor) will be used and dosing is according to standard institutional practice

SUMMARY:
This study aims to confirm non-inferiority of the BioFreedom™ Drug Coated Stent to the Gazelle™ Bare Metal Stent arm of the Leaders Free study (NCT01623180) in high bleeding risk patients.

DETAILED DESCRIPTION:
In this study all patients will receive the BioFreedom™ Drug Coated Stent and one month of Dual Anti Platelet Therapy

ELIGIBILITY:
Inclusion Criteria:

Any indication for percutaneous coronary intervention with stent placement (PCI-S) in patients deemed at high risk for bleeding and candidates for 1 month dual anti-platelet therapy (DAPT). This includes candidates with stable angina, silent ischemia, acute coronary syndrome (STEMI and non-STEMI), non-native lesions and in-stent restenosis. Patients must provide written informed consent.

Reasons of unsuitability for > 1 month dual antiplatelet treatment must include one or more of the following:

1. Adjunctive oral anticoagulation treatment planned to continue after PCI
2. Age ≥ 75 years old
3. Baseline Hgb <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to the index procedure)
4. Any prior intracerebral bleed
5. Any stroke in the last 12 months
6. Hospital admission for bleeding during the prior 12 months
7. Non skin cancer diagnosed or treated < 3 years, with a perceived increased risk for bleeding
8. Planned daily Nonsteroidal anti-inflammatory drugs (NSAID) (other than aspirin) or steroids for >30 days after PCI
9. Planned surgery that would require interruption of DAPT (within next 6 months)
10. Renal failure defined as: Creatinine clearance <40 ml/min
11. Thrombocytopenia (PLT <100,000/mm3)
12. Severe chronic liver disease defined as: patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice
13. Expected non-compliance to prolonged DAPT for other medical reasons

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Patients expected not to comply with 1 month DAPT
3. Patients requiring a planned staged PCI procedure more than one week after the index procedure
4. Procedure planned to require non-study stents, or stand-alone plain old balloon angioplasty (POBA) or stand-alone atherectomy
5. Active bleeding at the time of inclusion
6. Reference vessel diameter <2.25 - >4.0mm
7. Cardiogenic shock
8. Compliance with long-term single anti-platelet therapy unlikely
9. A known hypersensitivity or contraindication to aspirin, clopidogrel (or prasugrel, or ticagrelor if applicable), stainless steel, zinc, Biolimus A9™ or a sensitivity to contrast media, which cannot be adequately pre-medicated
10. PCI during the previous 12 months for a lesion other than the target lesion of the index procedure
11. Participation in another clinical trial (12 months after index procedure)
12. Patients with a life expectancy of < 12 months
13. Patients under judicial protection, tutorship or curatorship (for France only)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1203 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The composite of cardiac death and myocardial infarction at twelve months | 12 months
The incidence of clinically driven target lesion revascularization at twelve months | 12 months

SECONDARY OUTCOMES:
The composite of cardiac death and myocardial infarction | 1, 2, and 6 months and 2 and 3 years
The incidence of clinically driven target lesion revascularization | 1, 2, and 6 months and 2 and 3 years
The composite of cardiac death, myocardial infarction and stent thrombosis | 1, 2, and 6 months and 1, 2, and 3 years
Bleeding per Bleeding Academic Research Consortium (BARC) Criteria | 1, 2, and 6 months and 1, 2, and 3 years
Cardiac Death | 1, 2, and 6 months and 1, 2, and 3 years
Myocardial Infarction | 1, 2, and 6 months and 1, 2, and 3 years
Stent Thrombosis per Academic Research Consortium (ARC) Definition | 1, 2, and 6 months and 1, 2, and 3 years
Urgent target lesion revascularization | 1, 2, and 6 months and 1, 2, and 3 years
Clinically driven target lesion revascularization at time points other than primary endpoint | followed for all target lesion revascularizations, up to 3 years
Clinically driven target vessel revascularization | 1, 2, and 6 months and 1, 2, and 3 years
All cause mortality | 1, 2, and 6 months and 1, 2, and 3 years
Primary endpoints, in patients with at least 1 lesion treated with a trial stent of 3mm or less in nominal diameter | 1, 2, and 6 months and 1, 2, and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Leon, Study Chair — Cardiovascular Research Foundation, New York; Mitchell Krucoff, Principal Investigator — Duke University; Philip Urban, Principal Investigator — Hôpital de la Tour
Locations (66):
- United States (39):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Tri-Lakes Research, Hot Springs, Arkansas
  - Scripps Health, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Jacksonville, Jacksonville, Florida
  - Velella Research, Sarasota, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - North Georgia Heart Foundation, Gainesville, Georgia
  - St. Luke's Idaho Cardiology Associates, Boise, Idaho
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - St. Vincent Heart Center, Indianapolis, Indiana
  - Jewish and St. Mary's Hospital, Louisville, Kentucky
  - Lahey Clinic, Burlington, Massachusetts
  - McLaren Bay Region, Bay City, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - University of Buffalo, Buffalo, New York
  - Weill Cornell Medical College-New York Presbyterian, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Genesis Healthcare System, Zanesville, Ohio
  - Penn State - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Berks Cardiologists, Ltd., Reading, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Chattanooga Heart Institute, Chattanooga, Tennessee
  - Tennova Healthcare-Turkey Creek Medical Center, Knoxville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Providence Health Center, Waco, Texas
  - Carilion Clinic, Roanoke, Virginia
- Canada (11):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - The University of Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'université de Montréal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
  - CIUSSS de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Rigshospitalet Copenhagen University Hospital, Copenhagen, Denmark
- France (8):
  - Clinique Axium, Aix-en-Provence
  - Service de Cardiologie Interventionnelle - Pôle Santé République, Clermont-Ferrand
  - Clinique de Fontaine, Fontaine-lès-Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital Privé Jacques Cartier ICPS, Massy
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - Clinique Saint Hilaire, Rouen
  - CHU Toulouse Rangeuil, Toulouse
- Germany (2):
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Herzzentrum Leipzig GmbH, Leipzig
- Italy (2):
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera San Camillo Forlanini, Rome
- United Kingdom (3):
  - Royal Bournemouth Hospital, Dorset Heart Centre, Bournemouth
  - Craigavon Cardiac Centre, Craigavon
  - Golden Jubilee National Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
The emphasis in all scientific publications and presentations will be placed on the 1-year endpoint

REFERENCES:
- [Derived] Eberli FR, Oldroyd KG, Urban P, Krucoff MW, Morice MC, Tanguay JF, Leon MB, Brunel P, Maillard L, Lipiecki J, Cook S, Berland J, Hovasse T, Carrie D, Schutte D, Sadozai Slama S, Garot P. Clinical outcomes with thin versus thick strut polymer-free biolimus-coated stents at 3 years. Open Heart. 2024 Jun 18;11(1):e002679. doi: 10.1136/openhrt-2024-002679. PMID 38890129
- [Derived] Campos CM, Mehran R, Capodanno D, Owen R, Windecker S, Varenne O, Stone GW, Valgimigli M, Hajjar LA, Kalil Filho R, Oldroyd K, Morice MC, Urban P, Abizaid A. Risk Burden of Cancer in Patients Treated With Abbreviated Dual Antiplatelet Therapy After PCI: Analysis of Multicenter Controlled High-Bleeding Risk Trials. Circ Cardiovasc Interv. 2024 Apr;17(4):e013000. doi: 10.1161/CIRCINTERVENTIONS.122.013000. Epub 2024 Apr 16. PMID 38626080
- [Derived] Mehran R, Chandrasekhar J, Urban P, Lang IM, Windhoevel U, Spaulding C, Copt S, Stoll HP, Morice MC; LEADERS FREE Investigators. Sex-Based Outcomes in Patients With a High Bleeding Risk After Percutaneous Coronary Intervention and 1-Month Dual Antiplatelet Therapy: A Secondary Analysis of the LEADERS FREE Randomized Clinical Trial. JAMA Cardiol. 2020 Aug 1;5(8):939-947. doi: 10.1001/jamacardio.2020.0285. PMID 32432718